CLINICAL TRIAL: NCT02206737
Title: The Effects of Electronic Cigarettes on the Microcirculation of the Hand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CW14025
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Hand Injuries; Elective Hand Surgery
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- E-Cigarette (Experimental): 3 doses of e-cigarette to be given No nicotine Low dose nicotine High dose nicotine
  Interventions: Device: No nicotine e-cigarette; Device: Low dose nicotine e-cigarette; Device: High dose nicotine e-cigarette

INTERVENTIONS:
Device: No nicotine e-cigarette
Device: Low dose nicotine e-cigarette
Device: High dose nicotine e-cigarette

SUMMARY:
Cigarette smoking is associated with poor wound healing and worse results after hand surgery. Nicotine and cigarette smoke has been shown to affect blood flow in blood vessels in the hand.

Patients are increasingly using electronic cigarettes (e-cigarettes) as a method of quitting smoking. E-cigarettes consist of a replaceable nicotine cartridge, a heating element and a battery source. They are able to deliver vaporised nicotine in the absence of other ingredients found in normal cigarettes such as tar and carbon monoxide.

Although e-cigarettes lack a lot of the harmful ingredients of regular cigarettes, nicotine still has toxic effects on the body. Nicotine causes the release of chemicals within the body that act to reduce blood flow in small blood vessels of the hand.

E-cigarettes remain a controversial topic among healthcare professionals due to the lack of research surrounding them. A recently published literature review identified only three significant studies into the effects of smoking e-cigarettes. All of these studies showed the harmful effects of e-cigarettes on the lungs but to date, there is no published research investigating the effects of e-cigarettes on the blood flow within the small blood vessels of the hand.

Currently, we advise patients to quit smoking after they sustain a hand injury to improve healing and recent research suggests that patients should be advised to quit smoking 4 weeks before routine hand surgery. However, there is no guidance on whether we should also advice patients to refrain from using e-cigarettes for this time period.

Our aims are to answer the following questions:

1. Do electronic cigarettes have any effect on the blood flow in the hand?
2. Do we need to give cessation advice to patients with hand injuries who smoke electronic cigarettes?

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18-65yrs
* Volunteers with no co-morbidities
* Volunteers with no history of oral infections

Exclusion Criteria:

* Volunteers with ongoing co-morbidities requiring medical treatment
* Volunteers with a history of oral infections e.g Herpes Simplex Virus
* Volunteers who lack capacity to consent to the study
* Volunteers who are currently on nicotine replacement therapy
* Volunteers who have had use of a cigarette or nicotine containing product within 4 hours of beginning the study
* Volunteers who have previously quit smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Microcirculation after smoking different doses of electronic cigarettes | 2 hours
  Microcirculation prior to any intervention Microcirculation following inhalation of the e-cigarette with no nicotine cartridge installed (0-30 minutes) Microcirculation following inhalation of the e-cigarette with a low dose nicotine cartridge installed (0-30 minutes) Microcirculation following inhalation of the e-cigarette with a high dose nicotine cartridge installed (0-30 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster Hospital, London, London, United Kingdom

REFERENCES:
- [Background] Wei DH, Strauch RJ. Smoking and hand surgery. J Hand Surg Am. 2013 Jan;38(1):176-9; quiz 179. doi: 10.1016/j.jhsa.2012.08.018. Epub 2012 Nov 7. No abstract available. PMID 23141048
- [Background] Fischer-Rasokat U, Spyridopoulos I, Walter J, Honold J, Zeiher AM, Fichtlscherer S. Microvascular dysfunction and pulse wave reflection characterize different vascular pathologies in patients at cardiovascular risk. Vasa. 2012 May;41(3):192-9. doi: 10.1024/0301-1526/a000185. PMID 22565620
- [Background] Petschke FT, Engelhardt TO, Ulmer H, Piza-Katzer H. [Effect of cigarette smoking on skin perfusion of the hand]. Chirurg. 2006 Nov;77(11):1022-6. doi: 10.1007/s00104-006-1216-1. German. PMID 16896901
- [Background] van Adrichem LN, Hovius SE, van Strik R, van der Meulen JC. Acute effects of cigarette smoking on microcirculation of the thumb. Br J Plast Surg. 1992 Jan;45(1):9-11. doi: 10.1016/0007-1226(92)90106-8. PMID 1737221
- [Background] Bullen C, Howe C, Laugesen M, McRobbie H, Parag V, Williman J, Walker N. Electronic cigarettes for smoking cessation: a randomised controlled trial. Lancet. 2013 Nov 16;382(9905):1629-37. doi: 10.1016/S0140-6736(13)61842-5. Epub 2013 Sep 9. PMID 24029165
- [Background] Palazzolo DL. Electronic cigarettes and vaping: a new challenge in clinical medicine and public health. A literature review. Front Public Health. 2013 Nov 18;1:56. doi: 10.3389/fpubh.2013.00056. PMID 24350225